CLINICAL TRIAL: NCT05394662
Title: Safety and Effectiveness of Juveena™ Hydrogel System Following Transcervical Gynecologic Procedures (TCGP) At High-Risk for Intrauterine Adhesions: A Multicenter Randomized Controlled Subject and Evaluator Blinded Pivotal Study
Brief Title: Safety and Effectiveness of Juveena™ Hydrogel System Following TCGP At High-Risk for Intrauterine Adhesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rejoni Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REJ-CT-0003
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Intervention Model Description: Juveena Hydrogel vs No Hydrogel
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects won't be told which group they were assigned. Primary outcome reviewed by blinded independent central review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcervical Gynecological Procedure + Juveena Hydrogel (Experimental): Transcervical Gynecological Procedure + Juveena Hydrogel
  Interventions: Device: Juveena Hydrogel System
- Transcervical Gynecological Procedure alone (standard of care) (No Intervention): Transcervical Gynecological Procedure alone (standard of care)

INTERVENTIONS:
Device: Juveena Hydrogel System — Application of a novel hydrogel immediately following the transcervical procedure
  Arms: Transcervical Gynecological Procedure + Juveena Hydrogel

SUMMARY:
This study is to determine whether intrauterine instillation of Juveena hydrogel following adhesiogenic hysteroscopic procedures (TCGP + Juveena) can safely and effectively reduce the incidence and severity of intrauterine adhesions (IUA) compared to TCGP alone.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled subject and evaluator-blinded pivotal study to investigate the safety and effectiveness of the Juveena Hydrogel System when used to reduce the occurrence of IUA in women undergoing TCGPs associated with a high prevalence of post-procedural IUA (i.e., adhesiolysis for moderate to severe adhesions or myomectomy of multiple or large myoma). A second look hysteroscopy (SLH) will be performed at the Week 8 visit to evaluate the presence and severity of IUA.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal
2. Candidate for one of the following hysteroscopic procedures:

   1. Adhesiolysis of moderate to severe adhesions confirmed hysteroscopically
   2. Hysteroscopic Myomectomy confirmed via imaging in subjects with symptomatic disease
3. Subject agrees to all protocol requirements including returning for specified visits within intervals identified within this protocol.
4. Subject is willing to undergo an SLH at the Week 8 visit.
5. Subject agrees to abstain from sexual intercourse or use a reliable form of barrier contraception following the study procedure through the Week 8 visit.
6. Subject has signed the IRB/EC approved informed consent

Exclusion Criteria:

1. Postmenopausal
2. IUD present at time of TCGP (unless removed before or during procedure)
3. Past history of endometrial cancer or atypical endometrial hyperplasia (endometrial intraepithelial neoplasia).
4. Planned intrauterine interventions post-TCGP through the Week 8 visit.
5. Recent intrauterine surgery within 6 weeks before the planned study procedure.
6. Pregnant (positive pregnancy test) or lactating.
7. Pregnancy within the last 6 weeks prior to the planned study procedure for a trimester loss (≤13 weeks gestation) within 3 months of planned study procedure for all other pregnancies.
8. Active sexually transmitted infection (i.e., positive testing for gonorrhea/chlamydia), or genital or urinary tract infection at the time of procedure (e.g., cervicitis, vaginitis, endometritis, salpingitis, or cystitis) or other active and/or systemic infection.
9. Use of systemic corticosteroids within 1 week of study procedure.
10. Treated with long-acting injectable hormone/hormone implant that would still be active at the time of the TCGP.
11. Known allergy to FD&C No.1 dye or polyethylene glycol (PEG).
12. Known clotting defects or bleeding disorders.
13. Any other general health or mental condition that in the opinion of the investigator could represent an increased risk for the subject, affect the primary outcomes of this study and/or impact the subject's ability to comply with protocol requirements.
14. Participating or considering participation in a clinical trial of another investigational drug or device during this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Freedom from intrauterine adhesions (IUA) | 8 weeks
  Incidence of No IUA at second look hysteroscopy (SLH)

SECONDARY OUTCOMES:
Severity of IUA | 8 weeks
  Severity of IUA classified according to March criteria at SLH
Freedom of IUA with superiority margin of 5% over control at IUA | 8 weeks
  Incidence of No IUA with superiority margin of 5% over control

CONTACTS AND LOCATIONS:
Overall Officials: Ian Feldberg, Study Director — Rejoni Inc.
Locations (15):
- United States (15):
  - Arizona Gynecology Consultants, Phoenix, Arizona
  - UCSF Center for Reproductive Health, San Francisco, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Dr. Charles Miller and Associates, Park Ridge, Illinois
  - Cypress Medical Research Center, Wichita, Kansas
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Boston IVF, Waltham, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Duke Universtiy Health System, Morrisville, North Carolina
  - University Hospitals Landerbrook, Mayfield Heights, Ohio
  - Prisma Health, Greensville Memorial Hospital, Greenville, South Carolina
  - The University of Texas at Austin Dept of Womens' Health, Austin, Texas
  - Texas Fertility Center, Austin, Texas
  - Aspire Houston Fertility Institute, Houston, Texas
  - Generations Fertility Care, Middleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No